CLINICAL TRIAL: NCT02881788
Title: Minnesota Healthy Brain Initiative
Status: Completed | Type: Observational
Sponsor: Hennepin Healthcare Research Institute (Other)
Collaborators: Hennepin County Medical Center, Minneapolis (Other)
Responsible Party: Sponsor
Other Study IDs: HSR 16-4185
Record Dates: First submitted 2016-08-24; First posted 2016-08-29 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Cognitive Ability, General

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year

GROUPS / COHORTS (3):
- Traumatic Brain injury: There will be no intervention necessary. We will analyze the eyetracking data from subjects who have sustained a traumatic brain injury. We are hoping to find patterns that may indicate a TBI in the data we collect.
- Non-Traumatic Brain injury: There will be no intervention necessary. We will analyze the eyetracking data from subjects who have sustained a non-trauma related brain injury. We are hoping to find patterns that we may compare this data to subjects who have sustained a TBI as well as healthy controls.
- Control: There will be no intervention necessary. We will analyze the eyetracking data from subjects who have not recently sustained any brain injury. We are hoping to find patterns that we may compare this data to subjects who have sustained a TBI as well as subjects who have had a non-trauma related brain injury.

SUMMARY:
Minnesota Healthy Brain Initiative will be an ongoing project that aims to increase awareness regarding brain health and its maintenance as well as increasing awareness of the impact of alcohol on brain function. In the immediate future, we hope to obtain data from a non-injured normative, diverse population represented by the state fair patrons.

DETAILED DESCRIPTION:
We hypothesize that a non-invasive 30-minute test, requiring a subject to complete questionnaires and watch images on a TV screen, will yield information relevant to both diagnosis and prognosis of neurological state. To clarify, these tests will not produce information that would involve a diagnostic finding for the participants. We will measure eye movements under a range of visual conditions, including saccades, fixations, smooth pursuit, scan paths and optico-kinetic nystagmus

After receiving proper introduction and signing the proper consent forms, the subject will receive instructions to carry out cognitive assessments and answer verbal questionnaires. The subject will also undergo eye tracking. In order to validate the data collected by our eye-trackers, we may ask the subject to complete a non-invasive vision assessment and a breathalyzer assessment. Due to the nature of the breathalyzer assessment, we have decided not to administer the breathalyzer assessment to subjects who are under the age of 21 and/or pregnant. We also refuse to disclose the results of the breathalyzer assessment to the subject since the data will be collected only for research purposes. Subjects' eye movements will be tracked binocularly at a fixed distance from a computer monitor over a brief time period. The visual stimuli will be video clips appropriate for a general or pediatric audience. If at any point the subject becomes uncomfortable, the procedure will be aborted and can be resumed at a later time.

ELIGIBILITY:
Inclusion Criteria:

Males and Females Ages 4-100 All racial and ethnic origins will have an opportunity to participate

Exclusion Criteria:

Blind in one or both eyes Unable to open eyes Unable to detect light in either eye

Ages: 4 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Since we hope to gather a normative distribution, all subjects interested in participating in the study will be considered.
Sampling Method: Non-Probability Sample
Enrollment: 690 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Eyetracking | 0-1 yr
  The subject will complete a non-invasive eye tracking assessment. Our camera will follow the movement of their eye to assess the patterns made.

CONTACTS AND LOCATIONS:
Overall Officials: Uzma Samadani, MD, PHD, Principal Investigator — Hennepin County Medical Center, Minneapolis; Thomas Bergman, MD, Principal Investigator — Hennepin County Medical Center, Minneapolis